CLINICAL TRIAL: NCT06436651
Title: Evaluation of the Effectiveness of Digital Storytelling Method in Symptom Method in Children With Oncological Problems
Brief Title: Digital Storytelling in Symptom Management Pediatric Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Birgul Erdogan, Research Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E.795978
Record Dates: First submitted 2024-03-29; First posted 2024-05-31 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-06

CONDITIONS: Child, Only; Cancer; Symptoms and Signs; Narration
Keywords: child; cancer; nursing; symptom management; digital storytelling
MeSH Terms: conditions — Neoplasms; Signs and Symptoms; Narration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Children's group where digital storytelling method was applied and stories were created
  Interventions: Other: Digital Storytelling
- Control group (Other): Children's group where the stories of children in the initiative group will be watched
  Interventions: Other: Digital Storytelling

INTERVENTIONS:
Other: Digital Storytelling — 4 stages of digital storytelling will be implemented.

SUMMARY:
The aim of this clinical study is to evaluate the effectiveness of the digital storytelling method in symptom management in children diagnosed with oncology. It will also provide information about children's experiences with Digital Storytelling and the use of the method. The main questions it aims to answer are:

* Is there a difference between the anxiety scores of children who applied the Digital Storytelling Method and those who did not?
* Is there a difference between the fatigue scores of children who applied the Digital Storytelling Method and those who did not?
* Is there a difference between the nausea scores of children who applied the Digital Storytelling Method and those who did not?
* Is there a difference between the pain scores of children who applied and did not apply the Digital Storytelling Method?

Participants:

Complete the first stage data forms. Visit the clinic every 7-15 days for the digital storytelling process, which consists of 4 stages. After the storytelling process is completed, have a process evaluation meeting with the researcher.

DETAILED DESCRIPTION:
Participants; Enterprise Group,

1. Interview (Week 1); Meeting the child, conducting a qualitative interview for needs analysis and introducing the forms
2. Interview (Week 2); Finding a digital story topic
3. Interview (Week 3); Writing a story on the specified topic
4. Interview (Week 4); Converting the story into digital form
5. Interview (Week 5); Showing the created story
6. Interview (Week 6); Conducting a qualitative interview regarding the digital storytelling process.

Each meeting will be held in 1-week periods. Primary outcome tools will be applied as pretest and posttest once in the 1st and 6th interviews, and twice in the other interviews.

Control Group;

1. Interview (Week 1); Meeting the child, introducing and applying the forms
2. Interview (Week 6); Conducting a qualitative interview regarding the digital storytelling process. Showing the videos prepared by the children in the initiative group. Application of primary outcome tools.

ELIGIBILITY:
Inclusion Criteria:

* 7-18 years old,
* Having received at least 1 cure of treatment,
* Completed the induction phase and is in the consolidation phase,
* Children who and their parents agree to participate in the study.

Exclusion Criteria:

* who cannot speak Turkish,
* Having a secondary chronic disease
* Having a second disease that will affect the cognitive process,
* Children/adolescents who cannot complete the 4 stages of the digital storytelling process.
* Children/adolescents who cannot complete the 4 stages of the digital storytelling process.
* Children/adolescents who take a break of more than 3 weeks between storytelling processes.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2024-01-13 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory for Children | It will be used in the 1st and 6th interviews with the child (1st week-6th week).
  It will be used to evaluate children's state anxiety.
Visual Analogue Scale for Fatigue | It will be applied in all interviews with the child (6 interviews), before and after the interview. It will be applied 12 times in 6 weeks.
  It is a single-item scale used to determine the intensity of fatigue in patients. The patient is asked to score his or her fatigue on a scale of 0-10. 0 means no fatigue, while 10 is considered a lot of fatigue.
The Baxter Retching Faces Scale | It will be applied in all interviews with the child (6 interviews), before and after the interview. It will be applied 12 times in 6 weeks.
  The scale is applied to children/adolescents in the 7-18 age group. There are a total of six items in the scale, ranging from no force to vomiting, and six facial expressions indicating each item. While the scale can be used by asking the child to choose the face that best suits him/her, the cartoon can also be shown and evaluated through observation. The average application time of the scale is 2 minutes and scores are given between 0-10. Using 0 as 'no nausea' and 10 as 'vomiting'
Wong-Baker FACES pain rating scale (WB-FACES) | It will be applied in all interviews with the child (6 interviews), before and after the interview. It will be applied 12 times in 6 weeks.
  This scale is used to diagnose pain in children aged 3-18. This scale has six faces representing increasing pain intensity from zero to five from left to right. The far left face has a smiling expression, indicating a pain-free state, while the far right face has a crying expression, corresponding to the most severe pain. Six facial expressions are scored from left to right on a scale of 0 to 10 points (0 points = very happy/no pain, 10 points = most severe pain). As the score from the scale increases, pain tolerance decreases, and as the score decreases, tolerance increases. The child is told to choose the face that best expresses his or her emotions.

SECONDARY OUTCOMES:
SSPedi: Symptom Screening Scale in Pediatric Patients | It will be used in the 1st and 6th interviews with the child (1st week-6th week).
  The screening tool includes 15 symptoms that evaluate the symptoms children have experienced in the last two days. Each symptom is evaluated with a 5-point Likert-type scoring system, and the score range varies between 0-60. Higher scores indicate that the number of symptoms and the discomfort they cause increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Universıty, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No